CLINICAL TRIAL: NCT01240239
Title: Comparison of Telemedicine Evaluation to Standard Evaluation Methods for Pre-Anesthesia Consultation
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Richard Applegate, MD, Loma Linda University
Other Study IDs: 59305
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: ENT Patients Scheduled for Surgery
Keywords: Pre anesthesia consultation; telemedicine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- telephone group: The telephone group must be healthy adults scheduled for an ENT surgery.
- telemedicine group: This group if qualified will randomly be chosen to be in the telemedicine group.
- pre-anesthesia consultation: This will be the group that will be randomized to the pre-anesthesia clinic.

SUMMARY:
The purpose of the study is to evaluate different methods of pre-anesthesia consultation, with the aim of improving the day of surgery experience for the patient. In this study, we will use a telephone consultation, an in-person consultation, and a telemedicine consultation, which involves television cameras and monitors that allow live two-way communication for the pre-anesthesia consultation. The reason for this study is to evaluate the use of telemedicine for the pre-anesthesia consultation. Patients and anesthesiologists have been highly satisfied in previous studies using pre-anesthesia telemedicine consultation. In this study, we will examine a larger group of patients, as previous studies have studied smaller groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 89 who are scheduled for otolaryngologic procedures and pre-anesthesia consultation.

Exclusion Criteria:

Lack of consent; inability to understand English-

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects scheduled for ENT surgery.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Comparison Of Telemedicine Evaluation To Standard Evaluation Methods For Pre-Anesthesia Consultation | about 1 month
  Primary outcomes include surgical cancellation rate, delays the day of surgery secondary to inadequate pre-op evaluation, adequacy of the airway, respiratory, and cardiovascular exams, and intra-op and post-op complications. Patient data will include age, gender, ASA Physical Status and type of surgery. The length of the PACE appointment and the number of days prior to surgery the PACE appointment was conducted will be noted. Patient satisfaction with the will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Orange Tree Lane Otolaryngology Offices, Redlands, California, United States

REFERENCES:
- [Derived] Applegate RL 2nd, Gildea B, Patchin R, Rook JL, Wolford B, Nyirady J, Dawes TA, Faltys J, Ramsingh DS, Stier G. Telemedicine pre-anesthesia evaluation: a randomized pilot trial. Telemed J E Health. 2013 Mar;19(3):211-6. doi: 10.1089/tmj.2012.0132. Epub 2013 Feb 5. PMID 23384334